CLINICAL TRIAL: NCT03529526
Title: An Open-Label, Multi-center, Dose-Escalation Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetics and Immunogenicity of KN046 in Subjects With Advanced Solid Tumors
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Antitumor Activity of KN046 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alphamab (Australia) Co Pty Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN046-AUS-001
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: This is a dose-escalation trial, all participants will receive treatment with KN046. Participants enrolled in this trial may receive one of the following doses dependent upon time of enrolment into the study.
  Cohort 1: 0.3 mg/kg Cohort 2: 1 mg/kg Cohort 3: 3 mg/kg Cohort 4: 5 mg/kg Cohort 5: 10 mg/kg
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN046 (Experimental)
  Interventions: Drug: KN046

INTERVENTIONS:
Drug: KN046 — The modified phase I "3 + 3" study design was used in dose escalation from low dose to high dose to determine the MTD.Sequential assignment of Patient cohorts to one of five dose levels of KN046: 0.3 mg/kg,1 mg/kg,3 mg/kg,5 mg/kg,10 mg/kg.

SUMMARY:
This is an open-label, multicenter, dose-escalation phase I study to assess the safety, tolerability and preliminary efficacy of KN046 in participants with all advanced solid tumors who are not able to have current standard anti-tumor therapies. The purpose of this study is to determine the maximum tolerated dose (MTD) or a biological effective dose (BED), to characterise the safety, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of KN046 as a single agent in adult participants with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the informed consent form prior to the conduct of any study related procedures that are required during the screening period and are not considered part of standard of care.
2. Subjects must have histologic or cytologic confirmed Advanced solid tumors.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Adequate organ function within 3 weeks prior to initial treatment.
5. Ability to comply with treatment, procedures and PK sample collection and the required study follow-up procedures.
6. Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
7. Female patients must have a negative serum or urine pregnancy test
8. Female patients must not be breastfeeding.

Exclusion Criteria:

1. Subjects with brain metastases or leptomeningeal are excluded.
2. Concurrent enrollment in another clinical study, unless in a follow-up period or the study is an observational or non-interventional study.
3. Any kind of immunotherapy within 6 weeks of the first dose of study treatment.
4. Prior systemic cytotoxic chemotherapy, other anticancer drugs or growth factor within 28 days of the first dose of study treatment, or any investigational agents within 5 half-lives of the product.
5. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the 1st dose of study treatment, or have an anticipated need for major surgery during the study.
6. Palliative radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the 1st dose of study treatment.
7. Prior treatment or with sequential monotherapy with anti-CTLA-4 and anti-PD-1/PD-L agents.
8. Patients who have received monotherapy with PD-L1 / PD-1, CTLA4 or other antibodies and had intolerable toxicity or required steroids to manage toxicity.
9. History of autoimmune or inflammatory disorders.
10. A current or prior use of immunosuppressive medication within 14 days of the 1st dose of study treatment.
11. Suspected latent tuberculosis infection, confirmed by Mantoux test and a chest x-ray.
12. Any unresolved toxicity NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
13. Any factors that increase the risk of QT (ECG interval measured from the onset of the QRS complex to the end of the T wave) interval corrected for heart rate (QTc) prolongation or risk of arrhythmic events (e.g., heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age) or mean QTc>470 msec.
14. Positive blood screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus 1/2 antibody (HIV 1/2 Ab).
15. History of severe allergic reactions to any unknown allergens or to parenteral administered recombinant protein product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-05-21 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) | During the first cycle (4 weeks) of treatment.
  An DLT is defined as a ≥Grade 3 drug-related adverse event occurring within the first cycle (28 days) of dosing (excluding tumor flare causing local pain at sites of known or suspected tumor, localized rash, or a transient ≤Grade 3 infusion reaction) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of KN046，up to 2 years.
  An AE is defined as any untoward medical occurrence in a participant administered KN046 and/or pharmaceutical product(s) temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Objective response rate (ORR) | From first dose of KN046 through 90 days after last dose of KN046, up to 2 years.
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Duration of response (DoR) | up to 2 years.
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | From first dose of KN046 through 90 days after last dose of KN046, up to 2 years.
  Progression-free survival is defined as the time from the start of treatment with KN046 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Clinical benefit rate (CBR) | From first dose of KN046 through 90 days after last dose of KN046, up to 2 years.
  Clinical benefit rate is defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD) to KN046 intervention.
Area under the curve (AUC) of KN046 | From first dose of KN046 through 90 days after last dose of KN046, up to 9 months.
  The endpoints for assessment of PK of KN046 include serum concentrations of KN046 at different timepoints after KN046 administration.
Maximum observed concentration (Cmax) of KN046 | From first dose of KN046 through 90 days after last dose of KN046, up to 9 months.
  The endpoints for assessment of PK of KN046 include serum concentrations of KN046 at different timepoints after KN046 administration.
Minimum observed plasma concentration (Ctrough) of KN046 at steady state | From first dose of KN046 through 90 days after last dose of KN046, up to 9 months.
  The endpoints for assessment of PK of KN046 include serum concentrations of KN046 at different timepoints after KN046 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | Assessed before KN046 infusion in Cycle 1, 2, 3, 4, 5, 6 and at the mandatory Safety Follow-up Visit, maxium up to 2 years.
  The immunogenicity of KN046 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Number of subjects who develop detectable neutralizing ADA (NADA) | Assessed before KN046 infusion in Cycle 1, 2, 3, 4, 5, 6 and at the mandatory Safety Follow-up Visit, maxium up to 2 years.
  The neutralizing ADA will be assessed by summarizing the number of subjects who develop detectable neutralizing ADA .

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Cancer Care, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No